CLINICAL TRIAL: NCT01849848
Title: A Multicenter, Open-Label Phase II Study of SyB L-0501 in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Study of SyB L-0501 to Treat Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SymBio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011004
Record Dates: First submitted 2013-04-17; First posted 2013-05-09 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-02-06 (Estimated); Status verified 2015-01

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

ARMS (1):
- SyB L-0501 (Experimental)
  Interventions: Drug: SyB L-0501

INTERVENTIONS:
Drug: SyB L-0501 — The administration of SyB L-0501 at 90 mg/m^2/day by 60-minute intravenous infusion for 2 consecutive days followed by 26 days of monitoring. This is considered to be one cycle and may be repeated up to 6 times. Dose reduction or discontinuation is permitted from the second cycle as necessary according to adverse events and the results of monitoring during the previous cycle.

SUMMARY:
The purpose of this study is to determine the antitumor efficacy and safety of bendamustine (SyB L-0501: 90 mg/m^2/day) for a maximum of 6 cycles (1 cycle: intravenous administration for 2 consecutive days and 26-day observation period) in patients with relapsed/refractory multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed with multiple myeloma on the basis of the response criteria of the International Myeloma Working Group (IMWG) and confirmed to meet one or more of the following criteria:

   (definition of progression according to the IMWG response criteria)
   * 25% or more increase compared to baseline for the following values

     * Serum M-protein level (however, the absolute value is 0.5 g/dL or higher)
     * Urine M-protein level (however, absolute value is 200 mg/24 hours or higher)
     * For lesions without measurable serum or urine M-protein values. involved/uninvolved free light chain (FLC) ratio (however, absolute value is 10 mg/dL or higher)
   * Clear appearance of new bone lesions or soft tissue plasmacytoma or apparent growth in size of current bone lesions or soft tissue plasmacytoma
   * Appearance of hypercalcemia (corrected calcium level ≥ 11.5 mg/dL and if determined to be caused solely by myelomas)
2. Patients with measurable lesions (meets at least one of the following two criteria

   * Serum M-protein [Immunoglobulin G (IgG)≥ 1.0 g/dL, Immunoglobulin A (IgA) ≥ 0.5 g/dL, Immunoglobulin D (IgD) ≥ 0.1 g/dL)
   * Urine M-protein ≥ 200 mg/24 hours
3. Patients who meet either one of the following items for all prior chemotherapy using proteasome inhibitors, Immunomodulatory Drugs (IMiDs) (thalidomide or lenalidomide) or alkylating agents.

   * No response*
   * Relapse/recurrence after response*
   * Intolerance
   * Not applicable (reason can be confirmed in the source document) because of predicted aggravation of complications (neurotoxicity, etc.) * Patients whose disease has progressed based on the IMWG response criteria after receiving the most recent therapy
4. Patients who have undergone a washout period of more than 3 weeks after the end of the previous therapy and determined not to be under the effect of previous treatment (antitumor effectiveness).
5. Patients who are expected to survive for at least 3 months
6. Patients aged from 20 to 79 years at the time of interim registration
7. Performance Status (P.S.) of 0 to 125. However, P.S. 2 due to pain from lytic bone lesions is acceptable
8. Patients with adequately maintained organ functions (e.g., bone marrow, heart, lung, liver, and kidney functions)

   * Neutrophil count:≥ 1,500 /mm^3
   * Platelet count:≥ 75,000 /mm^3
   * Albumin:≥ 2.5 g /dL
   * Aspartate aminotransferase (AST) Glutamic oxaloacetic transaminase (GOT): < than 3.0 times the upper limit of normal range for the site
   * Alanine aminotransferase (ALT) Glutamic pyruvic transaminase (GPT): < than 3.0 times the upper limit of normal range for the site
   * Total bilirubin: < than 1.5 times the upper limit of normal range for the site
   * Serum creatinine: < than 3.0 times the upper limit of normal range for the site
   * Partial pressure of O2 (PaO2) ≥ 65 mmHg
   * No abnormalities which require treatment are detected on ECG
   * Left ventricular ejection fraction (LVEF)(echocardiography): ≥ 55%
9. Patients who have provided written consent for participation in this study

Exclusion Criteria:

1. Patients with apparent infections (including viral infections)
2. Patients with serious complications (hepatic or renal dysfunction, etc.)
3. Patients with complications or medical history of serious cardiac disease (e.g., myocardial infarction, ischemic heart disease) within 2 years of the date of interim registration or patients with arrhythmias that require treatment
4. Patients with serious gastrointestinal symptoms (e.g., severe nausea, vomiting, or diarrhea)
5. Patients positive for Hepatitis B surface (HBs) antigen, Hepatitis C virus (HCV) antibody, or HIV antibody
6. Patients with serious bleeding tendencies (e.g., disseminated intravascular coagulation: DIC)
7. Patients with, or confirmed in the past to have had, interstitial pneumonia, pulmonary fibrosis, or pulmonary emphysema which requires treatment.
8. Patients with a complication of apparent cardiac amyloidosis
9. Patients with infiltration to the central nervous system (CNS) or patients with clinical symptoms of suspected infiltration to the CNS,
10. Patients with active multiple primary cancer
11. Patients with, or confirmed in the past to have had, autoimmune hemolytic anemia
12. Patients who have received this investigational product in the past
13. Patients who have received allogeneic stem cell transplants in the past. (patients who have received autologous stem cell transplantation are acceptable)
14. Patients who received cytokine preparations such as erythropoietin or granulocyte colony stimulating factor (G-CSF) or blood transfusions within 1 week prior to the examination conducted before interim registration for this study
15. Patients who received other investigational products or unapproved medications within 3 months before interim registration for this study
16. Patients with prior allergies to medications that are similar to this investigational product (e.g., alkylating agents, or purine-nucleoside derivatives) or mannitol
17. Patients with drug addiction, narcotics addiction, and/or alcohol dependency
18. Patients who are pregnant, who may possibly be pregnant, or lactating
19. Patients who do not agree to practice contraception for the following periods:

    Male: During investigational product administration and until 6 months after final administration Female: During investigational product administration and until 4 months after final administration
20. Patients otherwise judged by the investigator or sub-investigator to be unsuitable for inclusion in this study

Ages: 20 Years to 79 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Japan (14):
  - Chūōku
  - Fukuoka
  - Isehara
  - Kōtoku
  - Kyoto
  - Nagoya
  - Niigata
  - Okayama
  - Sapporo
  - Sendai
  - Shibukawa
  - Shibuya-ku
  - Tokushima
  - Utsunomiya

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SyB L-0501
Started | 17
Completed | 13
Not Completed | 4
Not completed — Physician Decision | 1
Not completed — Progression of the primary disease | 3

BASELINE CHARACTERISTICS:
Arm/Group | SyB L-0501
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (9.8)
Age, Customized [Number; unit: participants]
  20-29 years | 0
  30-39 years | 0
  40-49 years | 2
  50-59 years | 3
  60-69 years | 7
  70-79 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 12
Subtype of myeloma [Number; unit: participants] — One participant could carry multiple subtypes of myeloma.
  participants
    Immunoglobulin G | 10
    Immunoglobulin A | 6
    Immunoglobulin D | 0
    Bence Jones type | 8
    κ | 13
    λ | 4
Prior therapy [Number; unit: participants]
  Absent | 0
  Present | 17
  Proteasome inhibitor | 17
  IMIDs | 16
  Alkylating agent | 17
  Other | 11
Performance status [Number; unit: participants] — The criteria of Eastern Cooperative Oncology Group (ECOG) performance status are shown below.
  0: Fully active, able to carry on all pre-disease performance without restriction , 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work , 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours
  participants
    0 | 7
    1 | 8
    2 | 2
Clinical disease stage (International Staging System) [Number; unit: participants] — The criteria of clinical disease stage (International Staging System) are shown below.
  stage I: Serum β2-microglobulin < 3.5 mg/L plus serum albumin ≥ 3.5 g/dL, stage II: neither stage I nor III , stage III: Serum β2-microglobulin ≥ 5.5 mg/L
  participants
    I | 3
    II | 11
    III | 3
Medical history [Number; unit: participants]
  Absent | 10
  Present | 7
Accompanying symptoms of the primary disease [Number; unit: participants]
  Absent | 1
  Present | 16
Complication [Number; unit: participants] — A complication is a disease or condition that arises as a result of multiple myeloma.
  participants
    Absent | 0
    Present | 17
Serum β2 microglobulin [Mean (Standard Deviation); unit: mg/L] | 4.03 (1.59)
Height [Mean (Standard Deviation); unit: cm] | 159.05 (9.95)
Body weight [Mean (Standard Deviation); unit: kg] | 56.86 (10.06)
Body surface area [Mean (Standard Deviation); unit: m^2] | 1.576 (0.181)

OUTCOME MEASURES:

1. Primary Outcome: Response Rate [Stringent CR (sCR)+Complete Response (CR)+Very Good PR (VGPR)+Partial Response (PR)]Based on International Myeloma Working Group (IMWG) Criteria
Description: The criteria for sCR, CR, VGPR, and PR based on IMWG are shown below.
  sCR: Fulfills CR criteria as well as all of the following conditions
  * Normal free light chain (FLC) ratio(κ/λ)
  * Disappearance of clonal cells in bone marrow by immunohistochemistry or immunofluorescence
  CR: Fulfills all of the following criteria
  * Negative immunofixation of serum and urine M-protein
  * <5% plasma cells in bone marrow
  * Disappearance of any soft tissue plasmacytoma
  VGPR: Fulfills at least one of the following criteria
  * Serum and urine M-protein detectable by immunofixation but not electrophoresis
  * ≥90% reduction in serum M-protein and 24-hour M-protein excretion amount in urine <0.1 g/24 hour
  PR: Fulfills the following criteria
  * ≥50% reduction in serum M-protein, and ≥90% reduction in urine M-protein, urine M-protein excretion amount is reduced to < 0.2 g/24hours
Time Frame: up to around 44 weeks
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 17
percentage of paticipants | 0 [0.0 to 19.5]

2. Secondary Outcome: Response Rate (sCR+CR) Based on IMWG Criteria
Time Frame: up to around 44 weeks
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 17
percentage of paticipants | 0 [0.0 to 19.5]

3. Secondary Outcome: Complete Response (CR) Based on the Blade Criteria
Description: The criteria for CR based on the Blade are shown below.
  CR requires all of the followings:
  1. Absence of the original monoclonal paraprotein in serum and urine by immunofixation, maintained for a minimum of 6 weeks
  2. <5% plasma cells in a bone marrow aspirate and also on trephine bone biopsy
  3. No increase in size or number of lytic bone lesions
  4. Disappearance of soft tissue plasmacytomas
Time Frame: up to around 44 weeks
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 17
percentage of paticipants | 0 [0.0 to 19.5]

4. Secondary Outcome: Response Rate (CR+PR) Based on the Blade Criteria
Description: The criteria for PR based on the Blade are shown below.
  PR requires 1. or all of the others:
  1. Some, but not all, of the criteria for CR are fulfilled
  2. ≥50% reduction in the level of the serum monoclonal paraprotein, maintained for a minimum of 6 weeks
  3. Reduction in 24 h urinary light chain excretion either by ≥90% or to <200 mg, maintained for a minimum of 6 weeks
  4. For patients with non-secretory myeloma only, ≥50% reduction in plasma cells in a bone marrow aspirate and on trephine biopsy
  5. ≥50% reduction in the size of soft tissue plasmacytomas
  6. No increase in size or number of lytic bone lesions
Time Frame: up to around 44 weeks
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 17
percentage of paticipants | 0 [0.0 to 19.5]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: Using the registration date as the start date, PFS with relapse/recurrence or progression, and death regardless of the cause as events are to be summarized using the Kaplan-Meier estimator and the 50% point according to the Greenwood's formula and the 95% confidence interval are to be calculated.
Time Frame: up to around 44 weeks
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | SyB L-0501
Number analyzed (Participants) | 17
Days | 92.0 [33.0 to 243.0]

6. Secondary Outcome: Time to Treatment Failure (TTF)
Description: Using the registration date as the start date, TTF with relapse/recurrence or progression, death regardless of the cause, and early discontinuation of treatment as events are to be summarized using the Kaplan-Meier estimator and the 50% point according to the Greenwood's formula and 95% confidence interval are to be calculated.
Time Frame: up to around 44 weeks
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | SyB L-0501
Number analyzed (Participants) | 17
Days | 71.0 [33.0 to 243.0]

7. Secondary Outcome: Duration of Response (DOR)
Description: From initial response (PR or higher), DOR with relapse/recurrence or progression, and death, regardless of cause, as events, are to be summarized using the Kaplan-Meier estimator and the 50% point according to the Greenwood's formula and 95% confidence interval are to be calculated.
Time Frame: up to around 44 weeks
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | SyB L-0501
Number analyzed (Participants) | 17
Days | NA [NA to NA] — Because there was no subject judged as "PR" or higher in this study.

8. Secondary Outcome: Overall Survival (OS)
Description: Using the registration date as the start date, OS with death, regardless of the cause, as events, are to be summarized using the Kaplan-Meier estimator and the 50% point according to the Greenwood's formula and 95% confidence interval are to be calculated.
Time Frame: up to around 44 weeks
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | SyB L-0501
Number analyzed (Participants) | 17
Days | 243.0 [185.0 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

9. Secondary Outcome: Adverse Events
Description: All adverse events occurring during the administration of the investigational product are to be examined for safety by cross tabulation lists and tables of incidence from the viewpoint of relationship with the drug, disease severity and medicine treated group.
Time Frame: up to around 44 weeks
Measure: Number; unit: participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 17
participants
  Any adverse event | 17
  Adverse drug reaction | 17
  SAE | 4
  Death | 0
  Discontinuation due to adverse events | 1

10. Secondary Outcome: Number of Subjects With Abnormality (Grade ≥3) in Laboratory Test Values
Description: Abnormalities in laboratory test values in overall study period were analyzed. Severity of abnormalities were evaluated using Common Terminology Criteria for Adverse Events (CTCAE). grade 1 : mild, grade 2 : moderate, grade 3 : severe or medically significant but not immediately life-threatening grade, 4 : life threatening or disabling grade, 5 : death related to adverse event
Time Frame: up to around 44 weeks
Measure: Number; unit: participants
Arm/Group | SyB L-0501
Number analyzed (Participants) | 17
participants
  CD4 lymphocytes decreased | 13
  Electrocardiogram QT corrected interval prolonged | 1
  Investigations - Other, sodium decreased | 2
  Investigations - Other, potassium decreased | 1
  Investigations - Other, calcium increased | 1
  Investigations - Other, Haemoglobin decreased | 2
  Lymphocyte count decreased | 16
  Neutrophil count decreased | 11
  Platelet count decreased | 2
  Weight increased | 1
  White blood cell decreased | 12

11. Secondary Outcome: Number of Abnormalities (Grade ≥3) in Laboratory Test Values
Description: as for outcome 10
Time Frame: up to around 44 weeks
Measure: Number; unit: Events
Arm/Group | SyB L-0501
Number analyzed (Participants) | 17
Events
  CD4 lymphocytes decreased | 14
  Electrocardiogram QT corrected interval prolonged | 1
  Investigations - Other, sodium decreased | 2
  Investigations - Other, potassium decreased | 2
  Investigations - Other, calcium increased | 1
  Investigations - Other, Haemoglobin decreased | 2
  Lymphocyte count decreased | 33
  Neutrophil count decreased | 15
  Platelet count decreased | 3
  Weight increased | 1
  White blood cell decreased | 17

ADVERSE EVENTS:
Time Frame: up to around 44 weeks
Arm/Group | SyB L-0501
Serious Adverse Events (participants affected / at risk) | 4/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SyB L-0501 (N=17)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pneumonia (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SyB L-0501 (N=17)
Anaemia (Blood and lymphatic system disorders) | 7
Conjunctivitis (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 5
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Haemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 8
Proctalgia (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Dyschezia (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Gait disturbance (General disorders) | 1
Generalised oedema (General disorders) | 2
Injection site reaction (General disorders) | 4
Malaise (General disorders) | 4
Oedema peripheral (General disorders) | 4
Pyrexia (General disorders) | 3
Injection site vasculitis (General disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 2
Periodontitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 5
Blood albumin decreased (Investigations) | 2
Blood calcium increased (Investigations) | 2
Blood chloride decreased (Investigations) | 2
Blood creatinine increased (Investigations) | 3
Blood lactate dehydrogenase increased (Investigations) | 2
Blood potassium decreased (Investigations) | 2
Blood pressure decreased (Investigations) | 1
Blood sodium decreased (Investigations) | 3
Blood urea increased (Investigations) | 2
Blood uric acid decreased (Investigations) | 2
Blood uric acid increased (Investigations) | 1
C-reactive protein increased (Investigations) | 5
CD4 lymphocytes decreased (Investigations) | 13
Electrocardiogram QT prolonged (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 2
Blood urine present (Investigations) | 4
Haemoglobin decreased (Investigations) | 7
Lymphocyte count decreased (Investigations) | 16
Neutrophil count decreased (Investigations) | 16
Neutrophil count increased (Investigations) | 2
Platelet count decreased (Investigations) | 12
Protein total decreased (Investigations) | 1
Protein total increased (Investigations) | 1
Red blood cell count decreased (Investigations) | 5
Weight decreased (Investigations) | 6
Weight increased (Investigations) | 1
White blood cell count decreased (Investigations) | 17
White blood cell count increased (Investigations) | 2
Protein urine present (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Urine output decreased (Investigations) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 3
Renal failure (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 2
Tooth extraction (Surgical and medical procedures) | 1
Hypertension (Vascular disorders) | 2
Dysuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No